CLINICAL TRIAL: NCT03033654
Title: Two Consecutive Sunscreen Applications Optimize Sun Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ida M. Heerfordt, MD, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-1-2014-094
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Sun Protection
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Two Consecutive Sunscreen Applications
  Interventions: Other: Sunscreen, Actinica

INTERVENTIONS:
Other: Sunscreen, Actinica — Two Consecutive Sunscreen Applications

SUMMARY:
The investigators aim to investigate how much two consecutive applications of sunscreen before sun exposure can increase the quantities of sunscreen applied and decrease the skin area left without sunscreen compared to a single application. Volunteers wearing swimwear applied sunscreen in a laboratory environment twice and had pictures taken in black light before and after. As sunscreens absorb black light the darkness of the skin increased with increasing amounts of sunscreen applied. The investigators conducted a standard curve establishing a link between picture darkness and applied sunscreen quantity. Participants were asked to apply sunscreen the way they would normally do but two consecutive times. No other advice was given. The level of protection was determined by picture analysis as measurements of darkness of selected skin sites as well as the percentages of skin area left without sunscreen in different body regions and in total.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasians between older than 18

Exclusion Criteria:

* Suffering from a skin disease, were allergic to the content in sunscreen, were pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sun protection | The day of intervention. Sun protection will be assessed right after sunscreen application.
  Sun protection will be determined as sunscreen quantities applied in mg/cm^2 and areas of covered skin in percentage.

IPD SHARING:
Plan to Share IPD: No